CLINICAL TRIAL: NCT06470633
Title: To Evaluate the Efficacy and Safety of Adebrelimab Combined With Chemotherapy Neoadjuvant Therapy in Early or Local Advanced Breast Cancer After Induction Treatment of High-intensity Focused Ultrasound and Adebrelimab
Brief Title: To Evaluate the Efficacy of Adebrelimab Combined With Chemotherapy After HIFU Induction Neoadjuvant Therapy HR+/HER2- Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wenbin Zhou, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJMU- BC03
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; HR+/HER2- Breast Cancer
Keywords: HR+/HER2- early breast cancer; HIFU; Immunotherapy; Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU+Adebrelimab+Chemotherapy (Experimental): Induction phase: HIFU+Adebrelimab Neoadjuvant Therapy phase: Adebrelimab+ EC-T(Epirubicin + Cyclophosphamide → Docetaxel
  Interventions: Drug: Adebrelimab; Procedure: High Intensity Focused Ultrasoun（HIFU）; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab 1200mg iv q3w
  Other Names: PD-Li
Procedure: High Intensity Focused Ultrasoun（HIFU） — HIFU treatment at lesion site
Drug: Cyclophosphamide — 600mg/m2 iv q3w
Drug: Epirubicin — 90mg/m2 iv q3w
Drug: Docetaxel — 75mg/m2 iv q3w

SUMMARY:
To explore the efficacy and safety of adebrelimab combined with chemotherapy (epirubicin + cyclophosphamide →docetaxel) neoadjuvant therapy early HR+/HER2- breast cancer with high risk factors after the induction treatment of HIFU and adebrelimab.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 years who require a negative pregnancy test for premenopausal and perimenopausal patients and promise to take reliable contraceptive measures during treatment;
2. Histopathologically confirmed breast cancer patients who with hormone receptor- positive, which defined as estrogen receptor (ER) ≥ 1%, and/ or progesterone receptor (PR) ≥ 1%, and HER-2 (0 or +), or ++,but FISH is no amplification;
3. Tumor size ≥ 3cm, and histological grade is 3 (poorly differentiated);
4. Regardless of lymph node status, but without distant metastasis;
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, they have at least one evaluable target lesion;
6. ECOG PS score: 0 - 1;
7. New York Heart Association (NYHA) functional class I;
8. Electrocardiogram without myocardial ischemia, echocardiography LVEF > 55%, cardiac markers: cardiac troponin I (cTnI) and brain natriuretic peptide (BNP) test values within the normal range;
9. Normal major organ function, Meet the following criteria:

WBC ≥ 4.0 × 10 9/L,Neutrophil count (ANC) ≥ 1.5 × 10 9/L; platelet ≥ 100 × 10 9/L; hemoglobin ≥ 10 g/dL; serum creatinine ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) ≤ 2.5 × ULN; alanine aminotransferase (ALT) ≤ 2.5 × ULN; total bilirubin ≤ 1.5 × ULN; serum creatinine ≤ 1.5 × ULN; 9.The subject is able to understand the study procedures, voluntarily join the study, sign the informed consent form, have good compliance, and cooperate with the follow-up.

Exclusion Criteria:

1. Patients during pregnancy and lactation, women of childbearing age who refuse to take effective contraceptive measures during the study period; Patients with peripheral nervous system disorders caused by diseases or those with a history of significant mental disorders and central nervous system disorders;
2. Serious or uncontrolled infections that may affect the evaluation of study treatment or study results, including but not limited to: active hepatitis virus infection, human immunodeficiency virus (HIV) antibody positive, lung infection, etc.;
3. Known allergy to the active ingredients or other components of the study drug or surgical contraindications;
4. In addition to cured basal cell carcinoma of the skin and cured cervical carcinoma in situ, other cancers are disease-free for less than 5 years;
5. Severe liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, active gastrointestinal ulcers and other need treatment;
6. Need to receive other anti-tumor therapy (except ovarian function inhibitors) during neoadjuvant therapy as judged by the investigator;
7. Patients who are participating in other clinical trials within one month;
8. Patients with severe heart disease or discomfort, Expected intolerance to chemotherapy,Including, but not limited to: a. fatal arrhythmia or higher grade atrioventricular block (second-degree type 2 [Mobitz 2] atrioventricular block or third-degree atrioventricular block); b. unstable angina pectoris; c. clinically significant valvular heart disease; d. transmural myocardial infarction on electrocardiogram; e. uncontrolled hypertension;
9. Any other conditions that in the opinion of the investigator would make the patient inappropriate for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
tpCR | 6 months
  total pathologic complete response rate（lymph node and breast）

SECONDARY OUTCOMES:
bpCR | 6 months
  breast pathologic complete response rate

IPD SHARING:
Plan to Share IPD: No